CLINICAL TRIAL: NCT00002855
Title: A Phase 3 Trial of Androgen Ablation Alone vs. Chemo/Hormonal Therapy as Initial Treatment of Unresectable/Metastatic Adenocarcinoma of the Prostate
Brief Title: Chemotherapy Plus Hormone Therapy Versus Androgen Suppression in Treating Patients With Metastatic or Unresectable Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM95-231; P30CA016672 (NIH); MDA-DM-95231 (Other: UT MD Anderson Cancer Center); NCI-G96-1044; CDR0000065105 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Doxorubicin; Estramustine; Flutamide; Ketoconazole; nilutamide; Hydrocortisone; hydrocortisone acetate; hydrocortisone hemisuccinate; Vinblastine; Castration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Arm I: Medical or surgical castration followed by an anti-androgen therapy with either flutamide, bicalutamide, or nilutamide.
  Interventions: Drug: Bicalutamide; Drug: Flutamide; Drug: Nilutamide; Procedure: Conventional Surgery
- Arm II (Experimental): Arm II: Chemo/hormonal therapy for 3 x 8-week courses, followed by total androgen blockade. Each course consists of 6 weeks of cytotoxic therapy with doxorubicin, ketoconazole, vinblastine, and estramustine followed by 2 weeks rest. Maintained on hydrocortisone both during treatment and during rest.
  Interventions: Drug: Doxorubicin hydrochloride; Drug: Estramustine Phosphate Sodium; Drug: Ketoconazole; Drug: Therapeutic Hydrocortisone; Drug: Vinblastine

INTERVENTIONS:
Drug: Bicalutamide
  Other Names: Casodex
  Arms: Arm I
Drug: Doxorubicin hydrochloride
  Other Names: Adriamycin; Adriamycin PFS; Adriamycin RDF; Rubex
  Arms: Arm II
Drug: Estramustine Phosphate Sodium
  Other Names: Emcyt
  Arms: Arm II
Drug: Flutamide
  Other Names: Eulexin
  Arms: Arm I
Drug: Ketoconazole
  Other Names: Nizoral
  Arms: Arm II
Drug: Nilutamide
  Other Names: Anandron; Nilandron
  Arms: Arm I
Drug: Therapeutic Hydrocortisone
  Other Names: A-hydroCort; Cortef; Cortenema; Cortifoam; Hydrocortone; Solu-Cortef
  Arms: Arm II
Drug: Vinblastine
  Other Names: Velban
  Arms: Arm II
Procedure: Conventional Surgery — Surgical castration
  Other Names: Castration
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining hormone therapy with chemotherapy and androgen suppression may kill more tumor cells. It is not yet known which treatment regimen is more effective for prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy plus hormone therapy versus androgen suppression alone as initial therapy in patients with prostate cancer that is metastatic or that cannot be removed surgically.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical benefit, as measured by time to progression and overall survival, of chemo/hormonal therapy compared to androgen ablation alone, when given as the initial systemic treatment in patients with acinar adenocarcinoma of the prostate that is not amenable to local therapy.
* Validate the clinical significance of PSA criteria for progression.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients are treated with medical or surgical castration followed by an anti-androgen therapy with either flutamide, bicalutamide, or nilutamide.
* Arm II: Patients receive chemo/hormonal therapy for 3 eight week courses, followed by total androgen blockade. Each course consists of 6 weeks of cytotoxic therapy with doxorubicin, ketoconazole, vinblastine, and estramustine followed by 2 weeks of rest. These patients are also maintained on hydrocortisone both during treatment and during rest.

Patients in arm II have a long-term central venous access device inserted.

PROJECTED ACCRUAL: A total of 368 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven acinar adenocarcinoma of the prostate
* Metastatic or locally advanced disease that either is not appropriately treated with surgery or radiation, or has recurred following previous "definitive" local therapy
* No CNS metastases
* No histologic subtypes, such as pure ductal or any component of small cell carcinoma
* Elevated PSA (at least 1.0 ng/mL in patients with prior prostatectomy or 4.0 ng/mL in those with prostate in place)

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Zubrod 0-2

Life expectancy:

* At least 3 years

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Conjugated bilirubin no greater than 0.8 mg/dL or total bilirubin no greater than 1.5 mg/dL
* Transaminase no greater than 4 times upper limit of normal

Renal:

* Creatinine clearance at least 40 mL/min

Cardiovascular:

* No evidence of bifascicular block on EKG
* No evidence of active ischemia on EKG
* No prior history of transient ischemic attack
* No evidence of congestive heart failure

Other:

* No active peptic ulcer disease
* No regular use of antacid or H2 blockers
* No known or predicted achlorhydria
* No concurrent use of terfenadine, astemizole, omeprazole, or cisapride
* No second malignancy unless curatively treated
* No history of deep venous thrombosis
* No history of pulmonary embolism
* No serious co-morbidity
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior cytotoxic systemic therapy

Endocrine therapy:

* Prior androgen deprivation therapy allowed if given for no more than 6 months to downstage primary
* No androgen deprivation therapy within 1 year prior to study

Radiotherapy:

* No prior cytotoxic systemic therapy (including systemic strontium-89 irradiation)
* Prior definitive radiotherapy to the prostate and/or one metastatic site allowed
* At least 8 weeks since radiotherapy to the pelvis
* At least 3 weeks since radiotherapy to a single metastatic site

Surgery:

* Prior prostatectomy allowed

Other:

* No concurrent anti-anginal therapy or aggressive anticoagulants

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 1996-08; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Time to Progression | From baseline to post treatment (minimally 24+ weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Randall E. Millikan, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Millikan RE, Wen S, Pagliaro LC, Brown MA, Moomey B, Do KA, Logothetis CJ. Phase III trial of androgen ablation with or without three cycles of systemic chemotherapy for advanced prostate cancer. J Clin Oncol. 2008 Dec 20;26(36):5936-42. doi: 10.1200/JCO.2007.15.9830. Epub 2008 Nov 24. PMID 19029421
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org